CLINICAL TRIAL: NCT00734955
Title: An Optical Assay System for Intra Operative Assessment of Tumor Margins in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00007857; 1R01EB011574-01A1 (NIH)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: Partial Mastectomy; Lumpectomy; Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reduction Mammoplasty (Experimental): Patients undergoing reduction mammoplasty
  Interventions: Device: 49-channel optical spectrometer
- Mastectomy (Experimental): Patients undergoing mastectomy
  Interventions: Device: 49-channel optical spectrometer
- Lumpectomy (Experimental): Patients undergoing a lumpectomy
  Interventions: Device: 49-channel optical spectrometer

INTERVENTIONS:
Device: 49-channel optical spectrometer

SUMMARY:
Our objective is to develop a novel optical assay system for intra operative assessment of tumor margins in partial mastectomy or mastectomy specimens. Our group has previously shown that optical techniques can effectively discriminate between malignant and non-malignant breast tissues. We have also shown that data collection and processing from a single point on the tissue specimen requires less than 5 seconds. In addition, the technique is easily adaptable to provide sensing depths that are required for breast margin assessment. The goal of the work proposed in this protocol is to test the sensitivity and specificity of an optical assay system developed by our group, for intra operative assessment of breast tumor margins.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Breast Cancer

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2006-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Identification of the optical signatures of breast tissue. | Day of procedure
  The primary outcome measure of this study is to identify the optical signatures of normal and cancerous tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Nimmi Ramanujam, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States